CLINICAL TRIAL: NCT06473909
Title: An Exploratory Clinical Study on the Efficacy and Safety of Humanized CD25 Monoclonal Antibody Combined With Glucocorticoid in the First-line Treatment of Acute Graft-versus-host Disease (aGVHD) After Allo-HSCT
Brief Title: Combination of Steroid and Humanized CD25 Monoclonal Antibody as First-line Therapy for aGVHD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024017
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Acute Graft Versus Host Disease
Keywords: aGVHD; humanized CD25 monoclonal antibody; glucocorticoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: CD25 antibody combined glucocorticoid as first-line treatment

INTERVENTIONS:
Drug: CD25 antibody combined glucocorticoid as first-line treatment — CD25 antibody combined glucocorticoid as first-line treatment

SUMMARY:
The first-line treatment of acute graft-versus-host disease with humanized CD25 monoclonal antibody combined with glucocorticoid was used to study the remission rate of acute graft-versus-host disease, the cumulative incidence and remission rate of severe acute graft-versus-host disease, GVHD-free survival rate, all-cause mortality and quality of life evaluation, and safety evaluation for prevention programs.

ELIGIBILITY:
Inclusion Criteria:

* ( 1 ) Diagnosis of grade II to IV acute graft-versus-host disease after hematopoietic stem cell transplantation.

( 2 ) older than or equal to 18 years old. ( 3 ) Informed consent can be signed by themselves. ( 4 ) HIV negative, HBV, HCV negative. ( 5 ) Informed consent must be signed before the start of the study procedure. The informed consent must be signed by the patient himself or his immediate family. Considering the patient 's condition, if the patient 's signature is not conducive to the treatment of the disease, the informed consent will be signed by the legal guardian or the patient 's immediate family.

Exclusion Criteria:

* • (1) diagnosed as VOD/SOS.

  * (2) Uncontrolled infection at enrollment; requires mechanical ventilation or is hemodynamically unstable at the time of enrollment;
  * (3) has severe hepatic insufficiency (defined as Child-Pugh Class C; has serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 xthe upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN.
  * (4) has end-stage renal impairment with a creatinine clearance less than 10 mL/min.
  * (5) has both moderate hepatic insufficiency AND moderate renal insufficiency;
  * (6) has documented positive results for human immunodeficiency virus antibody (HIVAb), hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) within 90 days prior to enrollments;
  * (7) has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (e.g., lymphomas).
  * (8) Suffering from mental disorders or other conditions and unable to cooperate with the requirements of study treatment and monitoring;
  * (9) unable or unwilling to sign the consent form;
  * (10) patients with other special conditions assessed as unqualified by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The remission rate of aGVHD | 28 days

SECONDARY OUTCOMES:
Incidence rate of severe aGVHD | 24 weeks
overall survival | 24 weeks
infection rate | 24 weeks
relapse rate | 24 weeks
non-relapse mortality | 24 weeks

IPD SHARING:
Plan to Share IPD: No